CLINICAL TRIAL: NCT03193879
Title: Effects of Particulate Matter on the Lung Function and Acute Exacerbation of COPD and Asthma Patients--A Multi-center Cohort Study
Brief Title: Effects of Particulate Matter on the Pulmonary Function and Acute Exacerbation of COPD and Asthma
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Xinjiang Autonomous Region People 's Hospital (Unknown); Cangzhou Central Hospital (Other); Chengdu sixth People 's Hospital (Unknown); Chengde Central Hospital (Other Government); Beijing Fengtai Hospital (Unknown); The Affiliated Hospital of Medical College, Ningbo University (Other); Changzhi Medical College (Other); Beijing Boai Hospital (Other); Wuhu County Traditional Chinese Medicine Hospital (Other); The First People's Hospital of Jingzhou (Other); Fujian Provincial Hospital (Other); Harbin Zhongshan Asthma Hospital (Unknown); Rizhao Hospital of Chinese Traditional Medicine (Unknown); 3201 Hospital in Hanzhong (Other); Sir Run Run Shaw Hospital (Other); Chengdu Fifth People's Hospital (Other); First People 's Hospital of Changsha (Unknown); Chongqing Jiangjin Central Hospital (Unknown); the Affiliated hospital of Guilin medical university, China (Unknown); Jiangxi People 's Hospital (Unknown); Chinese People 's Liberation Army Navy Anqing Hospital (Unknown); The Affiliated Hospital of Inner Mongolia Medical University (Other); Yancheng Dafeng People 's Hospital (Unknown); ShuGuang Hospital (Other); The First Affiliated Hospital of the Fourth Military Medical University (Other); Taizhou Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Third Affiliated Hospital of Xinjiang Medical University (Other); First People 's Hospital of Kunming (Unknown); First People 's Hospital of Yunnan (Unknown); Pingxiang People 's Hospital (Unknown); Northern Jiangsu People 's Hospital (Unknown); Xiangya Hospital of Central South University (Other); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Second Hospital of Jilin University (Other); The Second Economic Hospital of Xinjiang Uygur Autonomous Region (Unknown); Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015CB553402
Record Dates: First submitted 2017-06-14; First posted 2017-06-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Pulmonary Function
Keywords: Pulmonary function; Particulate matter; COPD; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Biological specimens are preserved in serum, plasma, and leukocytes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COPD group: COPD patients
- Asthma group: Asthma patients
- Health group: Healthy volunteers

SUMMARY:
Particulate matter(PM) exposure has been shown to increase the morbidity and mobility of a variety of respiratory diseases, including COPD and asthma. This study focus on the effects of PM on the pulmonary function and acute exacerbation of COPD and asthma patients in China, where PM exposure is much heavier than the United States and European countries.

DETAILED DESCRIPTION:
Particulate matter(PM) exposure has been shown to increase the morbidity and mobility of a variety of respiratory diseases, including COPD and asthma. This study focus on the effects of PM on the pulmonary function and acute exacerbation of COPD and asthma patients in China, where PM exposure is much heavier than the United States and European countries. This study is an observational study which lasts 3 years. Primary outcome measures:Change in spirometry (FEV1) of COPD, asthma patients and healthy volunteers in response to different exposure doses of PM.

ELIGIBILITY:
Inclusion Criteria:

1. COPD patients: clinical manifestation of COPD; post bronchodilator FEV1/FVC<0.70.
2. Asthma patients: clinical manifestation of asthma; recurrent dyspnea; with or without wheezing; relief spontaneously or after using bronchodilators; FEV1/FVC<0.70,with positive bronchial reversible test.
3. Asthma combined with COPD (ACOS) patients: patients with ACOS are included in asthma group.
4. Healthy volunteers: No smoking history, or have quit smoking at least 5 years. Chest X-ray show no abnormality.
5. Information consent form should be signed before entering the study.

Exclusion Criteria:

1. The latest severe acute attack occurred within 4 weeks:

   1. Severe acute attack: status asthmaticus or acute exacerbation of COPD leading to consultation, emergency treatment，hospitalization, or glucocorticoid treatment（oral/i.v).
   2. Controllable non-hospitalized acute attack without glucocorticoid treatment(oral/i.v). COPD attack lasting less than 48h or asthma attack lasting less than 24h are not excluded.
2. Any history of acute/chronic respiratory diseases other than asthma and COPD, including lung cancer and pulmonary infection.
3. Plasma ALT or AST greater than 2 times of the upper normal limit; plasma Creatinine greater than 1.5 times of the upper normal limit.
4. Left heart insufficiency, or malignant arrhythmia.
5. HIV positive.
6. Acute cerebrovascular events within 3 months, including apoplexy, transient cerebral ischemia and acute coronary syndrome.
7. Uncured malignant tumors.
8. Addicted to drug or alcohol, or any history of psychiatric disorders.
9. Breastfeeding, pregnancy or planning to be pregnant.
10. Estimated lifetime less than 2 years due to underlying diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinic-based population
Sampling Method: Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Change in spirometry (FEV1) of COPD, asthma patients and healthy volunteers in response to different exposure doses of PM. | 2 years
  Spirometry will be assessed at baseline and through study completion, an average of 2 years.

SECONDARY OUTCOMES:
Change in morbidity of acute exacerbation in COPD and asthma patients in response to different exposure doses of PM. | 2 years
  Patients will be followed up through study completion, an average of 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided